CLINICAL TRIAL: NCT06668688
Title: Evaluation of the Naturalistic User Experience of the Website "ich Bin Alles @Schule" (i Am Everything @school) - an Information Platform for Educational Professionals on Depression and Mental Health in Childhood and Adolescence
Brief Title: Evaluation of the Naturalistic User Experience of the Website "ich Bin Alles @Schule" (i Am Everything @school)
Status: Recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Prof. Otto Beisheim Foundation (Other)
Responsible Party: Principal Investigator, Lisa Feldmann, Postdoctoral Researcher, LMU Klinikum
Other Study IDs: 24-0395-KB
Record Dates: First submitted 2024-10-24; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Depression; Depressive Disorder; Depression in Children; Depression in Adolescence
Keywords: depression; prevention; web-based; adolescents; mental health; school; user experience; acceptance; teachers
MeSH Terms: conditions — Depression; Depressive Disorder; Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 24-0395-KB: Naturalistic User Experience "ich bin alles @Schule"
  Interventions: Device: "ich bin alles @Schule" (i am everything @school; www.schule.ich-bin-alles.de)

INTERVENTIONS:
Device: "ich bin alles @Schule" (i am everything @school; www.schule.ich-bin-alles.de) — The web-based information platform for educational professionals "ich bin alles @Schule" (i am everything @school; www.schule.ich-bin-alles.de) on depression and mental health in childhood and adolescence was developed by the Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy at the LMU Munich Hospital together with the Prof. Otto Beisheim Foundation. The website is intended to provide low-threshold information about depression and mental health in the school context.

SUMMARY:
The aim of this study is to investigate the naturalistic user experience and acceptance of the German website "ich bin alles @Schule". This website for educational professionals offers information on depression and mental health of pupils. Another aim of this study is to determine whether the desired target groups of the website can be reached.

DETAILED DESCRIPTION:
Depressive disorders are among the most common psychiatric disorders in childhood and adolescence and yet often are unnoticed and not treated for a long time. Depressive disorders often begin in adolescence and young adulthood. School stress, caused by bullying experiences at school or high performance expectations from parents and teachers, has been identified as an important factor in the development of depressive disorders in students. School, as a central area of life for children and young people, is an important place for promoting pupils' mental health. The rising prevalence of depressive disorders among adolescence in recent years and the delayed start of interventions show a clear need for action in the everyday lives of adolescents. The Department of Child and Adolescent Psychiatry of the Hospital of the LMU Munich and the Beisheim Foundation launched the innovative digital information portal "Ich bin alles @Schule" (i am everything @school; www.schule.ich-bin-alles.de) in November 2023. "ich bin alles @Schule" is a German information platform that was developed for educational professionals and aims to provide low-threshold information about depression and mental health in the school context.

Due to the high relevance of comprehensively evaluating web-based information services on mental health and mental illness, the aim of this study is to use established methods to learn more about the visitors of "ich bin alles @Schule" and their user experience.

The aim of the study is a scientific evaluation of the naturalistic user experience of "Ich bin alles @Schule" users. For this purpose, an online questionnaire and the website analysis tool "Matomo" is applied. The study is intended to provide clues as to whether the "ich bin alles @Schule" information platform is a useful and trustworthy source of information for the target group. The information obtained is of central importance for potential adaptations and optimizations of the website. Another aim of this study is to determine whether we can actually reach the desired target group with our website. The results of the data collection also provide an important basis for future approaches aimed at school professionals about mental health issues and mental illness in a way that is appropriate for the target group.

ELIGIBILITY:
Inclusion Criteria:

* 40 seconds Website-use

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: users of the website "ich bin alles @Schule" (i am everything @school; www.schule.ich-bin-alles.de)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The characteristics of the people who are interested in "ich bin alles @Schule" (i.e. the users) | 40 seconds after Website-use
  Assessed via self-designed questionnaire
Perception of the users of website content | 40 seconds after Website-use
  Assessed via WEB-CLIC-S (Thielsch & Hirschfeld, 2021)
Perceived Website Usability | 40 seconds after Website-use
  Assessed via Perceived Website Usability - German (PWU-G; Flavián et al., 2006; Thielsch, 2008)
Visual Aesthetics of Website | 40 seconds after Website-use
  Assessed via Visual Aesthetics of Website Inventory - Short (VisAWI-S; Moshagen & Thielsch, 2013)
Intention to revisit the website | 40 seconds after Website-use
  Assessed via Scale assessing the intention to revisit the website (Moshagen & Thielsch, 2010)
Overall impression | 40 seconds after Website-use
  Assessed via a single item by Thielsch (2008)

SECONDARY OUTCOMES:
Specific data collected for "ich bin alles @Schule" with Matomo | two years (from website launch until anticipated stuy completion)
  Title of the pages accessed (page title)
Specific data collected for "ich bin alles @Schule" with Matomo | two years (from website launch until anticipated stuy completion)
  Location of the users: Country, region, city, approximate latitude and longitude (geolocation)
Specific data collected for "ich bin alles @Schule" with Matomo | two years (from website launch until anticipated stuy completion)
  Number of the website users
Specific data collected for "ich bin alles @Schule" with Matomo | two years (from website launch until anticipated stuy completion)
  How users accessed the website (e.g. Google search or Social Media link)
Specific data collected for "ich bin alles @Schule" with Matomo | two years (from website launch until anticipated stuy completion)
  How much time (seconds) users spend on the website

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Schulte-Körne, Prof. Dr., Study Director — Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, LMU University Hospital
Locations (1):
- LMU University Hospital (recruitment is conducted online), Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coppens E, Van Audenhove C, Iddi S, Arensman E, Gottlebe K, Koburger N, Coffey C, Gusmao R, Quintao S, Costa S, Szekely A, Hegerl U. Effectiveness of community facilitator training in improving knowledge, attitudes, and confidence in relation to depression and suicidal behavior: results of the OSPI-Europe intervention in four European countries. J Affect Disord. 2014 Aug;165:142-50. doi: 10.1016/j.jad.2014.04.052. Epub 2014 May 4. PMID 24882192
- [Background] Doll CM, Michel C, Rosen M, Osman N, Schimmelmann BG, Schultze-Lutter F. Predictors of help-seeking behaviour in people with mental health problems: a 3-year prospective community study. BMC Psychiatry. 2021 Sep 3;21(1):432. doi: 10.1186/s12888-021-03435-4. PMID 34479537
- [Background] Liao Y, Ameyaw MA, Liang C, Li W. Research on the Effect of Evidence-Based Intervention on Improving Students' Mental Health Literacy Led by Ordinary Teachers: A Meta-Analysis. Int J Environ Res Public Health. 2023 Jan 4;20(2):949. doi: 10.3390/ijerph20020949. PMID 36673704
- [Background] Thapar A, Eyre O, Patel V, Brent D. Depression in young people. Lancet. 2022 Aug 20;400(10352):617-631. doi: 10.1016/S0140-6736(22)01012-1. Epub 2022 Aug 5. PMID 35940184
- [Background] Thielsch, M. T., & Hirschfeld, G. (2021). Quick Assessment of Web Content Perceptions. International Journal of Human-Computer Interaction, 37(1), 68-80. https://doi.org/10.1080/10447318.2020.1805877
- [Background] Thielsch, M. T. (unter Mitarbeit von Salaschek, M.) (2017). Toolbox zur kontinuierlichen Website-Evaluation und Qualitätssicherung (Version 2.1). Arbeitsbericht, Köln: Bundeszentrale für gesundheitliche Aufklärung (BZgA). http://dx.doi.org/10.17623/BZGA:224-2.1
- [Background] Tong Y, Wang S, Cao L, Zhu D, Wang F, Xie F, Zhang X, Wang G, Su P. School dropouts related to mental disorders: A systematic review and meta-analysis. Asian J Psychiatr. 2023 Jul;85:103622. doi: 10.1016/j.ajp.2023.103622. Epub 2023 May 8. No abstract available. PMID 37172421
- [Background] Vieira MA, Gadelha AA, Moriyama TS, Bressan RA, Bordin IA. Evaluating the effectiveness of a training program that builds teachers' capability to identify and appropriately refer middle and high school students with mental health problems in Brazil: an exploratory study. BMC Public Health. 2014 Feb 28;14:210. doi: 10.1186/1471-2458-14-210. PMID 24580750
- [Background] Weist MD, Hoover SA, Daly BP, Short KH, Bruns EJ. Propelling the Global Advancement of School Mental Health. Clin Child Fam Psychol Rev. 2023 Dec;26(4):851-864. doi: 10.1007/s10567-023-00434-7. Epub 2023 May 29. PMID 37247024
- [Background] Flavián, C., Guinalíu, M., & Gurrea, R. (2006). The role played by perceived usability, satisfaction and consumer trust on website loyalty. Information & Management, 43(1), 1-14.
- [Background] Moshagen, M. & Thielsch, M. T. (2010). Facets of visual aesthetics. International Journal of Human Computer Studies, 68 (10), 689-709. http://dx.doi.org/10.1016/j.ijhcs.2010.05.006
- [Background] Moshagen, M. & Thielsch, M. T. (2013). A short version of the visual aesthetics of websites inventory. Behaviour & Information Technology, 32 (12), 1305-1311. http://dx.doi.org/10.1080/0144929X.2012.694910
- [Background] Thielsch, M. T. (2008). Ästhetik von Websites. Wahrnehmung von Ästhetik und deren Beziehung zu Inhalt, Usability und Persönlichkeitsmerkmalen. Münster: MV Wissenschaft.
- See also: German website "ich bin alles @Schule" Information portal on depression and mental health in children and young people for educational professionals — https://schule.ich-bin-alles.de/